CLINICAL TRIAL: NCT01467622
Title: Prospective, Non Randomized Investigator Initiated Multi-centre Trial on the Effects of Local Treatment Protocols on the Duration of Chest Tube Therapy Following Thoracic Surgery in Germany
Brief Title: Effects of Local Protocols on Duration of Chest Tube Therapy Following Thoracic Surgery
Status: Completed | Type: Observational
Sponsor: Schillerhoehe Hospital (Other)
Collaborators: Medela AG (Industry)
Responsible Party: Principal Investigator, Thorsten Walles, Prinicpal Investigator, Schillerhoehe Hospital
Other Study IDs: KSH-TCH-IIT-2009-1
Record Dates: First submitted 2011-10-30; First posted 2011-11-09 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Pulmonary Air Leak
Keywords: chest tube drainage; pulmonary air leak; lung resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study population: Patients undergoing elective pulmonary wedge resection, anatomic segmentectomy, or lobectomy.
  Interventions: Procedure: Chest tube removal

INTERVENTIONS:
Procedure: Chest tube removal — Chest tube removal on the basis of local recommendations for postoperative chest tube management

SUMMARY:
The effect of local chest-tube management protocols on the duration of chest-tube therapy following thoracic surgery was analyzed in four German specialized Thoracic Surgery Units. The primary study objective was the duration of chest tube therapy in postoperative patients.

DETAILED DESCRIPTION:
The management of chest tubes is probably one of the most critical aspects in patient care in thoracic surgery and defines the required length of postoperative hospital stay in the majority of patients. So far, no generally accepted recommendations exist for postoperative chest tube management to streamline the postoperative stay. Instead, decision making in most thoracic surgery units is based on team preferences and individual training rather than scientific data. Therefore, digital pleural drainage systems represent a useful tool to standardize existing intradepartmental protocols for chest tube management. However, for the development of generally accepted protocol-recommendations, the diverging interdepartmental treatment protocols have to be analyzed and compared for superiority. In this IIT, the effect of different chest tube management protocols on chest tube duration is analyzed in four German Thoracic Surgery units.

ELIGIBILITY:
Inclusion Criteria:

* age 18-85
* following pulmonary wedge resection, anatomic segmentectomy, or lobectomy

Exclusion Criteria:

* surgery for spontaneous pneumothorax (primary and secondary)
* surgery for pleural empyema
* present medication with corticoids, immunosuppressive drugs or platelet aggregation inhibitors other than Aspirin
* history of chemotherapy, radiotherapy of the chest, or previous ipsilateral thoracic surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing pulmonary resection at one of the four participating thoracic surgery specialist units
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2009-04; Primary Completion 2009-08 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
chest tube therapy duration | participants are followed for the duration of hospital stay, an expected average of 5 days
  number of days following thoracic surgery until chest tube was removed

SECONDARY OUTCOMES:
presence of pulmonary air leak | participants are followed for the duration of hospital stay, an expected average of 4 days
  number of days the Medela Thopaz device detected a pulmonary air leak following thoracic surgery

CONTACTS AND LOCATIONS:
Overall Officials: Albert Linder, MD, Study Director — Klinikum Bremen-Ost gGmbH; Thorsten Walles, MD, Principal Investigator — Schillerhoehe Hospital; Josef Wolf, Study Chair — Medela GmbH & Co. Handels KG
Locations (4):
- Germany (4):
  - Evangelische Lungenklinik Berlin, Berlin
  - Klinikum Bremen-Ost gGmbH, Bremen
  - Klinik Schillerhoehe, Gerlingen
  - Katholisches Klinikum Koblenz, Koblenz

REFERENCES:
- [Result] Linder A, Ertner C, Steger V, Messerschmidt A, Merk J, Cregan I, Timm J, Walles T. Postoperative chest tube management: snapshot of German diversity. Interact Cardiovasc Thorac Surg. 2012 Oct;15(4):622-6. doi: 10.1093/icvts/ivs270. Epub 2012 Jun 29. PMID 22753431